CLINICAL TRIAL: NCT03201003
Title: AR101 Trial in Europe Measuring Oral Immunotherapy Success in Peanut Allergic Children (ARTEMIS)
Brief Title: ARTEMIS Peanut Allergy In Children
Acronym: ARTEMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC010
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Peanut Allergy
Keywords: AR101; Characterized Peanut Allergen; CPNA (Characterized Peanut Allergen); OIT (oral immunotherapy); Peanut Allergy; Peanut-Allergic Children; Desensitization; ARTEMIS; Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Severe combined immunodeficiency with sensitivity to ionizing radiation; Hypersensitivity | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AR101 (Active Comparator): AR101 powder provided in capsules & sachets
  Interventions: Biological: AR101 powder provided in capsules & sachets
- Placebo (Placebo Comparator): Placebo powder provided in capsules & sachets
  Interventions: Other: Placebo powder provided in capsules & sachets

INTERVENTIONS:
Biological: AR101 powder provided in capsules & sachets — Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol
  Arms: AR101
Other: Placebo powder provided in capsules & sachets — Study product formulated to contain only inactive ingredients for use as defined in the protocol
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of AR101 through oral immunotherapy (OIT) in peanut-allergic children.

DETAILED DESCRIPTION:
This is a European, multicenter, double-blind, randomized, placebo-controlled 2-arm study of the efficacy and safety of AR101 in peanut-allergic children.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 4 to 17 years, inclusive
* Clinical history of allergy to peanuts
* Serum SPT ≥ 3 mm greater than control and/or psIgE ≥ 0.35 kUa/L
* Dose limiting symptoms after consuming a single dose of peanut protein ≤ 300 mg
* Written informed consent from the subject's parent/guardian
* Written assent from the subject as appropriate (per local regulatory requirements)
* Use of effective birth control by sexually active female subjects of childbearing potential

Key Exclusion Criteria:

* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* History of severe asthma (NHLBI criteria steps 5 or 6), or mild to moderate asthma (2007 NHLBI criteria steps 1-4) that is uncontrolled or difficult to control
* History of severe or life threatening episode of anaphylaxis or anaphylactic shock within 60 days of screening
* History of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD), symptoms of dysphagia or recurrent gastrointestinal symptoms of undiagnosed etiology
* History of a mast cell disorder, including mastocytosis, urticaria pigmentosa, chronic idiopathic or chronic physical urticaria beyond simple dermatographism (e.g., cold urticaria, cholinergic urticaria), and hereditary or idiopathic angioedema
* Any other condition that, in the opinion of the Investigator, precludes participation for reasons of safety

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Director — Aimmune Therapeutics
Locations (18):
- France (4):
  - Unité de dermatologie Pédiatrique, Hôpital Pellegrin-Enfants, place Amélie Raba-Léon, Bordeaux
  - Hopital Saint Vincent de Paul, Service d'Allergologie, Lille
  - Paediatric Allergy and Pulmonology Center, Jeanne de Flandre Hospital, Lille University Hospital, Lille
  - Service d'Allergologie Nouvel Hôpital Civil Hôpitaux Univesitaires de Strasbourg, Strasbourg
- Germany (2):
  - Charité Universitaetsmedizin Berlin, Klinik für Pädiatrie mit Schwerpunkt Pneumologie und Immunologie, Berlin
  - University of Frankfurt, Klinik für Kinder- und Jugendmedizin, Pädiatrische Allergologie, Pneumologie und Mukoviszidose, Frankfurt am Main
- Ireland (2):
  - UCC Dept. of Paediatrics and Child, Cork University Hospital, Cork
  - National Children's Research Centre, Our Lady's Children's Hospital Crumlin, Dublin
- Azienda Ospedaliera di Padova, Padua, Italy
- Spain (3):
  - Hospital General Universitario Gregorio Marañón, C/Manuel Esquerdo 46, Madrid
  - H. Infantil Universitario Niño Jesús, Servicio de Alergia, Madrid
  - Hospital Clinico San Carlos, Madrid Hospital Clinico San Carlos, Madrid
- Sachsska Children and Youth Hospital, Stockholm, Sweden
- United Kingdom (5):
  - James Paget University Hospital, Gorleston-on-Sea, Norfolk
  - Guy & St Thomas' Hospital, NHS Foundation Trust, London
  - St. Mary's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - University Hospitals Southampton Foundation NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blumchen K, Kleinheinz A, Klimek L, Beyer K, Anagnostou A, Vogelberg C, Butovas S, Ryan R, Norval D, Zeitler S, Du Toit G. Post hoc analysis examining symptom severity reduction and symptom absence during food challenges in individuals who underwent oral immunotherapy for peanut allergy: results from three trials. Allergy Asthma Clin Immunol. 2023 Mar 13;19(1):21. doi: 10.1186/s13223-023-00757-8. PMID 36915184
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504
- [Derived] Fernandez-Rivas M, Vereda A, Vickery BP, Sharma V, Nilsson C, Muraro A, Hourihane JO, DunnGalvin A, du Toit G, Blumchen K, Beyer K, Smith A, Ryan R, Adelman DC, Jones SM. Open-label follow-on study evaluating the efficacy, safety, and quality of life with extended daily oral immunotherapy in children with peanut allergy. Allergy. 2022 Mar;77(3):991-1003. doi: 10.1111/all.15027. Epub 2021 Sep 24. PMID 34320250
- [Derived] O'B Hourihane J, Beyer K, Abbas A, Fernandez-Rivas M, Turner PJ, Blumchen K, Nilsson C, Ibanez MD, Deschildre A, Muraro A, Sharma V, Erlewyn-Lajeunesse M, Zubeldia JM, De Blay F, Sauvage CD, Byrne A, Chapman J, Boralevi F, DunnGalvin A, O'Neill C, Norval D, Vereda A, Skeel B, Adelman DC, du Toit G. Efficacy and safety of oral immunotherapy with AR101 in European children with a peanut allergy (ARTEMIS): a multicentre, double-blind, randomised, placebo-controlled phase 3 trial. Lancet Child Adolesc Health. 2020 Oct;4(10):728-739. doi: 10.1016/S2352-4642(20)30234-0. Epub 2020 Jul 20. PMID 32702315

RESULTS

PARTICIPANT FLOW:
Groups:
- AR101: AR101 drug product was supplied in 2 presentations. These were pull-apart capsules containing 0.5, 1, 10, 20 and 100mg of peanut protein and sealed sachets containing 300mg of peanut protein.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
- Placebo: A placebo matching the AR101 drug product was supplied in 2 presentations. These were capsules matching the 0.5, 1, 10, 20 and 100mg peanut capsules but containing no peanut protein, and sealed sachets matching the peanut protein sachets but without any peanut protein. The capsules were used during the Initial Escalation and Up-dosing phases of the study, while the sachets were used during the Maintenance phase.
Period: Overall Study
Arm/Group | AR101 | Placebo
Started | 132 | 43
Completed | 106 | 40
Not Completed | 26 | 3
Not completed — Adverse Event | 14 | 1
Not completed — Other reasons | 5 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR101 | Placebo | Total
Number analyzed (Participants) | 132 | 43 | 175
Age, Customized [Count of Participants; unit: Participants]
  Children (4-11 years) | 97 | 30 | 127
  Adolescents (12-17 years) | 35 | 13 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 16 | 80
  Male | 68 | 27 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 119 | 39 | 158
  Unknown or Not Reported | 11 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 106 | 34 | 140
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 23 | 7 | 30
Region of Enrollment [Number; unit: participants]
  Sweden | 8 | 3 | 11
  Ireland | 20 | 6 | 26
  United Kingdom | 46 | 13 | 59
  Italy | 5 | 3 | 8
  France | 12 | 5 | 17
  Germany | 21 | 7 | 28
  Spain | 20 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Ages 4-17 Who Tolerated a Single Highest Dose of at Least 1000 mg in the Exit Oral Food Challenge.
Description: The proportion of subjects in the ITT population who achieve desensitization as determined by tolerating specified challenge doses of peanut protein with no more than mild symptoms at the Exit Oral Food Challenge.
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 132 | 43
Participants | 77 | 1
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference at 1000 mg; Test type: Superiority; p < 0.0001, Fisher Exact; Risk Difference (RD) = 56.0, 95% CI 2-sided [44.1 to 65.2]

2. Secondary Outcome: Proportion of Subjects Ages 4-17 Who Tolerated a Single Highest Dose of at Least 600 mg in the Exit Oral Food Challenge
Description: as for outcome 1
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 132 | 43
Participants | 90 | 4
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference at 600 mg; Test type: Superiority; p < 0.0001, Fisher Exact; Risk Difference (RD) = 58.9, 95% CI 2-sided [44.2 to 69.3]

3. Secondary Outcome: Proportion of Subjects Ages 4-17 Who Tolerated a Single Highest Dose of at Least 300 mg in the Exit Oral Food Challenge.
Description: as for outcome 1
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 132 | 43
Participants | 97 | 7
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference at 300 mg; Test type: Superiority; p < 0.0001, Fisher Exact; Risk Difference (RD) = 57.2, 95% CI 2-sided [41.2 to 69.1]

4. Secondary Outcome: Maximum Severity of Symptoms at Any Challenge Dose During the Peanut Exit Oral Food Challenge
Description: The maximum severity of symptoms on 4 levels: 0-None, 1-Mild, 2-Moderate, 3-Severe or higher (severe, life threatening, fatal) observed in the DBPCFC at any dose (1000 mg or lower)
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 132 | 43
Participants
  None | 47 | 0
  Mild | 55 | 16
  Moderate | 24 | 20
  Severe or higher | 6 | 7
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference in Maximum Severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel statistic (with equally spaced scores) stratified by country

ADVERSE EVENTS:
Time Frame: Approximately 9 months
Arm/Group | AR101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/132 | 2/43
Other Adverse Events (participants affected / at risk) | 130/132 | 42/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR101 (N=132) | Placebo (N=43)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Paracetamol and a combination hormone birth control medication. Unrelated to treatment.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR101 (N=132) | Placebo (N=43)
Flushing (Vascular disorders) | 15 (42) | 1 (3)
Systemic allergic reaction (Immune system disorders) | 16 (22) | 1 (2)
Seasonal allergy (Immune system disorders) | 10 (20) | 2 (2)
Pyrexia (General disorders) | 29 (41) | 14 (19)
Fatigue (General disorders) | 13 (36) | 5 (5)
Malaise (General disorders) | 8 (12) | 3 (3)
Chest discomfort (General disorders) | 7 (15) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 57 (659) | 8 (25)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 43 (157) | 7 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (166) | 24 (53)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 34 (89) | 10 (22)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 23 (63) | 8 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (40) | 3 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 22 (45) | 3 (8)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 10 (31) | 1 (8)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 11 (19) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 37 (99) | 12 (18)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 7 (37) | 2 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 3 (7)
Lymphadenopathy (Blood and lymphatic system disorders) | 8 (10) | 1 (1)
Headache (Nervous system disorders) | 46 (128) | 19 (65)
Dizziness (Nervous system disorders) | 4 (4) | 3 (3)
Eye pruritus (Eye disorders) | 24 (37) | 8 (12)
Eye swelling (Eye disorders) | 11 (18) | 3 (7)
Ear pain (Ear and labyrinth disorders) | 14 (21) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 4 (5) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 88 (835) | 19 (126)
Nausea (Gastrointestinal disorders) | 58 (437) | 11 (31)
Paraesthesia oral (Gastrointestinal disorders) | 52 (961) | 9 (49)
Vomiting (Gastrointestinal disorders) | 53 (120) | 10 (17)
Oral pruritus (Gastrointestinal disorders) | 28 (236) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 20 (112) | 4 (6)
Lip pruritus (Gastrointestinal disorders) | 16 (97) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 17 (120) | 2 (3)
Tongue pruritus (Gastrointestinal disorders) | 12 (133) | 5 (11)
Lip oedema (Gastrointestinal disorders) | 7 (20) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 16 (26) | 8 (19)
Abdominal pain upper (Gastrointestinal disorders) | 14 (44) | 5 (6)
Lip pain (Gastrointestinal disorders) | 7 (21) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 67 (300) | 14 (62)
Urticaria (Skin and subcutaneous tissue disorders) | 48 (156) | 9 (27)
Erythema (Skin and subcutaneous tissue disorders) | 34 (69) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 21 (38) | 8 (18)
Angioedema (Skin and subcutaneous tissue disorders) | 13 (87) | 4 (7)
Eczema (Skin and subcutaneous tissue disorders) | 12 (25) | 11 (18)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (5)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (15) | 1 (1)
Conjunctivitis (Infections and infestations) | 15 (31) | 5 (25)
Nasopharyngitis (Infections and infestations) | 44 (77) | 12 (21)
Rhinitis (Infections and infestations) | 20 (51) | 7 (17)
Viral infection (Infections and infestations) | 18 (24) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 17 (21) | 11 (12)
Gastroenteritis (Infections and infestations) | 12 (13) | 5 (6)
Gastroenteritis viral (Infections and infestations) | 7 (8) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (4) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03201003/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03201003/SAP_001.pdf